CLINICAL TRIAL: NCT00194805
Title: Telehealth for Diabetes Self-Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-5886-V03; 1K01NR008506-03 (NIH)
Record Dates: First submitted 2005-09-15; First posted 2005-09-19 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Diabetes; Aging
Keywords: Internet; Diabetes; Education; Social Support
MeSH Terms: conditions — Diabetes Mellitus | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Subjects randomized into the treatment group received the computer treatment
  Interventions: Behavioral: Telehealth for Diabetes Self Management; Other: Telehealth for Diabetes Self Management

INTERVENTIONS:
Behavioral: Telehealth for Diabetes Self Management
Other: Telehealth for Diabetes Self Management — Web based education format delivered for a six month period

SUMMARY:
This study will examine the feasibility and short and-long-term efficacy of a web-based telehealth intervention with community-dwelling older adults who have been diagnosed with type 2 diabetes. Effectiveness will be evaluated using multiple measures within three different domains: 1) physical (glycosylated hemoglobin [HbA1C], weight, and lipid levels); 2) behavioral (monitoring blood glucose levels, feet inspections, diet, and exercise frequency), and 3) psychosocial (depression, quality of life, social support, and adjustment to diabetes).

This is a randomized controlled trial of a web-based telehealth intervention designed to improve self-management behaviors in a group of community dwelling older diabetics. Two groups of participants will be recruited and randomized over a four-month period during years 01 and 02. Participants in the control group will receive standard diabetic care provided by their provider. Participants in the intervention group will receive computer training in the participant's home in how to access and utilize the web-based telehealth study webpage. The intervention will consist of a program designed and delivered via the Internet to improve the participants' diabetes self-management behaviors using behavioral and motivational strategies and cues to modify perceptions of self-efficacy and beliefs regarding the ability to affect the progress of the disease and change personal behavior.

DETAILED DESCRIPTION:
This one year study plans to enroll 62 individuals into two groups. One group will receive the standard diabetic care provided and the second group will receive the standard diabetic care and training on how to use a computer to access the Internet. Participant assignment into either group is random (like flipping a coin). Study procedures will include the completion of questionnaires; a blood pressure reading, weight and a finger prick to obtain a blood sample.

There will be a total of three visits. One visit will occur before the study starts and at a six-month interval during the study period. The time to complete the study procedures by the research staff is approximately 1 to 1½ hours.

1. Questionnaires: Participants will meet with a research staff person who will ask questions about dietary intake, exercise activity, blood glucose levels, feet inspections, past and current Internet activity, and psychosocial well-being (depression, quality of life, self-efficacy, social support, readiness to change, and adjustment to diabetes). The time estimated for completion is about 45 to 60 minutes.
2. Physiologic Measures: Participants will have their blood pressures taken, weight measured using a scale, and asked to provide 4-5 drops of blood from the fingertip to measure glycosylated hemoglobin (HbA1c), Cholesterol (HDL:LDL ratio) will be measured to evaluate improvement in short-and-long term (3 months to one year) management of diabetes.
3. Participants selected to participate in the computer/Internet study group will be contacted by research staff within one month to schedule a time to set-up the study computer equipment and receive computer training. Three 2 hour sessions of computer training over a three-week period in participants' homes will be scheduled. Participants will also be expected to participate in following Internet study procedures, available via the Internet from their homes.

   1. Maintaining a daily personal log of diabetes self care activities (blood sugar readings, diet, exercise, feet inspections, etc.)
   2. Participating in nurse led peer support question and answer chat sessions twice a month.

   d). Read and respond to e-mail sent from the study nurse. e) Read health information on diabetes management, depression, and psychosocial well being that will be provided by the study nurse.

   Computer Training Training will be provided on how to use the computer, access the study web page resources, and participate in the nurse-led peer support group conference forum, use e-mail, and how to prepare and send a daily log of self-management activities (blood sugar monitoring, diet, feet inspections, and exercise). Training will also be provided on how to use the study web site's bulletin board, and the electronic prompt to verify completion of the weekly health reading assignment, and how to develop and post an action plan on-line.

   The amount of time for the above Internet activities will vary depending on participants' degree of interest in accessing the Internet resources provided. Approximately 1-4 hours per week or more will be needed to complete the Internet activities. Participants who are assigned to the intervention group who fail to respond to e-mail or to use any of the intervention resources for a one-week period will be contacted by telephone to determine the reason for not participating in the study activity (technical, knowledge deficit, medical, lack of ability, lack of interest, etc.).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Type 2 diabetes (American Diabetes Association criteria), i.e., fasting blood sugar levels of 126 mg/d or non-fasting levels of 200 mg/d when not taking glycemic control medication for diabetes
* diagnosed with diabetes for at least one year
* living in a non-institutional home in the community
* age 60 or older
* willing to be randomized
* able to read and write English or have an available caregiver or family member who can provide the necessary language translation.

Exclusion Criteria:

* moderate to severe cognitive impairment (less than 24 on the Mini Mental State Examination)
* severe vision impairment (greater than or equal to 9 on the Functional Vision Screening Scale);
* impairment of Activities of Daily Living (greater than 2 on Katz's Activities of Daily Living Scale);
* inability to hold and move objects; push buttons or use a trackball or a telephone;
* the presence of terminal debilitating medical conditions likely to result in death or severe disability prior to completion of the study;
* severe expressive or receptive communication impairment (inability to communicate will interfere with the administration of outcome measures), or
* no available phone-line or free electrical outlet

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2003-09; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
glycosylated hemoglobin (A1C) levels. | one year

SECONDARY OUTCOMES:
Study participants who receive the web-based telehealth intervention will have fewer depression symptoms and higher quality of life, social support, at post-test (short-term) than participants in the control group. | 1 year
Study participants who receive the web-based telehealth intervention will have fewer depression symptoms and higher quality of life, social support, at the 12 month (long-term) follow-up than participants in the control group. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Gail E Bond, Ph.D, Principal Investigator — University of Washington; Fredric Wolf, Ph.D, Study Chair — University of Washington; Martha Price, DNs, Study Director — University of Washington; Linda Teri, PhD, Study Chair — University of Washington; Jerry Palmer, Study Chair — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States